CLINICAL TRIAL: NCT06746961
Title: A Single-arm, Open-label, Multicenter Phase Ⅰb/Ⅱ Clinical Study of QL1706 (bispecific Antibody Targeting PD-1 and CLTA-4) in Combination with Lenvatinib in Second-line Therapy for Advanced Esophageal Squamous Cell Carcinoma After Disease Progression on Immune Checkpoint Blockades Therapy
Brief Title: Efficacy and Safety of QL1706 Plus Lenvatinib As 2nd Line Theapy in Patients with Metastatic Esophageal Carcinoma After Disease Progression on ICIs Therapy
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-EC-IIT-001
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: QL1706; lenvatinib; immune checkpoint blockades; esophageal squamous cell carcinoma; ESCC
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- QL1706 plus Lenvatinib (Experimental): QL1706 will be administrated at a dose of 5 mg/kg intravenously (IV), every 3 weeks, until progressive disease or intolerable or other reasons according to the criteria for termination of treatment. QL1706 will be administrated up to 2 year.
  Lenvatinib will be administrated at a dose of 8 mg or 12mg orally (PO) once daily (QD)
  Interventions: Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4); Drug: Lenvatinib

INTERVENTIONS:
Drug: QL1706 (bispecific antibody targeting PD-1 and CLTA-4) — 5mg/kg , iv, q3w
Drug: Lenvatinib — 8 mg or 12 mg QD via oral capsule
  Other Names: MK-7902; E7080; LENVIMA

SUMMARY:
The purpose of this study is to assess the efficacy and safety of QL1706 plus lenvatinib in second-line therapy for patients with metastatic esophageal squamous cell carcinoma after progression on immune checkpoint inhibitor therapy

ELIGIBILITY:
Inclusion Criteria:

1. Subjects participate voluntarily and sign informed consent.
2. 18-75 years, male or female.
3. Histologically or cytologically verified diagnosis of unresectable locally advanced or metastatic esophageal squamous cell carcinoma
4. Patients who have disease progression verified by imaging on standard first-line immunotherapy with anti-PD-1/PD-L1 antibodies
5. At least 1 measurable target lesion according to Response Evaluation in Solid Tumors (RECIST 1.1).
6. ECOG PS 0-1

Exclusion Criteria:

1. Presence of any active autoimmune disease or history of autoimmune disease (such as: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, nephritis, hyperthyroidism)
2. Those who are taking immunosuppressants or systemic hormonal therapy for immunosuppressive purposes (dose> 10 mg/day prednisone or other equivalent cortiremonial hormones) and are taking within 2 weeks before recruitment
3. Severe allergic reaction to other monoclonal antibodies
4. Those who terminated treatment due to related toxicity during anti-PD-1/PD-L1 antibody treatment
5. Prior treatment with bispecific anti-PD-1/CTLA-4 checkpoint blockades or VEGFR inhibitors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Phase Ib：Dose Limiting Toxicities (DLTs) and recommended phase 2 dose (PR2D) | up to ~21 days
  Hematologic DLTs are defined as:
  1. Grade 4 neutropenia lasting for ≥7 days
  2. febrile neutropenia not associated with the underlying disease,
  3. Grade 3 thrombocytopenia with bleeding, Grade ≥3 thrombocytopenia requiring platelet transfusion, Grade 4 thrombocytopenia, .
Phase II: Overall Survival (OS) in all participants | up to ~48 months
  OS is defined as the time from the first administration to death due to any cause.

SECONDARY OUTCOMES:
PFS | up to ~42 months
  PFS is defined as the time from the first administration to the first documented progressive disease (PD) per RECIST 1.1 by investigators or death due to any cause, whichever occurs first.
ORR | up to ~42 months
  ORR is defined as the percentage of participants with Complete Response or Partial Response per RECIST 1.1 assessed by the investigators.
DOR | up to ~42 months
  For participants who demonstrate a confirmed CR or PR, per RECIST 1.1 by the investigators, DOR is defined as the time from first documented evidence of CR or PR until PD or death.
Number of Participants With AEs | Up to ~53 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.